CLINICAL TRIAL: NCT01781026
Title: A Phase 2 Study of Neoadjuvant Vemurafenib in Melanoma Patients With Untreated Brain Metastases, Whose Tumors Harbor B-raf Mutations
Brief Title: Phase 2 Study of Neoadjuvant Vemurafenib in Melanoma Patients With Untreated Brain Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1208010666
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Results first posted 2015-04-02 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-01

CONDITIONS: Melanoma
Keywords: B-raf V600E; V600K mutation; metastatic melanoma
MeSH Terms: conditions — Melanoma | interventions — Vemurafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vemurafenib Administration (Experimental): Vemurafenib 960 mg orally, twice per day
  Interventions: Drug: Vemurafenib

INTERVENTIONS:
Drug: Vemurafenib — Single arm trial
  Other Names: Zelboraf / RO5185426

SUMMARY:
The purpose of this trial is to study the activity of vemurafenib in untreated melanoma brain metastases harboring B-Raf proto-oncogene, serine/threonine kinase (BRAF) mutations that are not amenable to stereotactic radiosurgery based on size, number of lesions or location, to measure cerebrospinal fluid (CSF) levels of vemurafenib as an indicator of central nervous system penetrance and to measure levels of vemurafenib in normal brain tissue and brain metastases in those in whom surgical management is feasible.

DETAILED DESCRIPTION:
This is a phase II single arm study. After establishing eligibility, including at least one lesion that is not amenable to immediate stereotactic radiosurgery (SRS) or surgical resection based on size or location OR more than four lesions, patients will begin therapy with vemurafenib at 960 mg PO BID continuous dosing. Any lesions deemed in need of and amenable to urgent local therapy will be treated prior to initiation of vemurafenib, provided that patients have at least one untreated evaluable lesion.

An MRI of the brain will be obtained after 4 weeks of vemurafenib therapy. If the CNS index lesion(s) are stable or shrinking, an additional 4 weeks of vemurafenib will be given with the goal of providing definitive local therapy at 8 weeks. If any lesion is growing after 4 weeks, depending on the size and concern for symptom evolution, the PIs can either continue vemurafenib for 4 additional weeks or provide definitive local or regional therapy at the 4 week mark in the form of surgery, Laser Induced Thermal Therapy (LITT), Stereotactic Radiosurgery (SRS) or Whole Brain Radiation Therapy (WBRT). If a lesion becomes symptomatic at any time, local therapy can be administered, and the patient can remain on study provided that there is an additional untreated brain metastasis. If the patient receives LITT or has surgical resection, biopsy samples will be sent to the sponsor for measurement of vemurafenib levels in tumor and normal brain parenchyma. Levels of pERK, as a surrogate for vemurafenib activity, will be measured in tumor samples. Vemurafenib will be held on the morning of radiation and restarted the following day. Vemurafenib dosing will not be held for surgery.

All patients will be asked to have a lumbar puncture after 4 weeks of vemurafenib therapy. The next MRI of the brain will be obtained at week 8 and then every 8 weeks, along with body CT or PET/CT scans.

If a patient is having overall shrinkage or stable disease in most CNS lesion(s), but if an individual cerebral metastases enlarges, local therapy can be done on study at any time if necessary. Patients will continue on vemurafenib until they have overall disease progression in either their CNS lesion(s) or in their systemic metastases as determined by modified MacDonald criteria (for cerebral lesion(s)) or RECIST criteria (for systemic disease), toxicities that preclude continuing the study drug, withdrawal from study, development of other severe illness, neurologic or systemic complications following local therapy to any lesion, termination of study, or death. Dose reductions for toxicities will be allowed.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven metastatic melanoma with the B-raf V600E or V600K mutations.
* Untreated brain metastases
* At least one cerebral metastasis that is not amenable to stereotactic radiosurgery (SRS) or surgical resection based on size or location OR four or more lesions
* Patients may be symptomatic at the time of enrollment, but after any necessary local therapy and/or corticosteroids, the patient should be asymptomatic when vemurafenib is initiated.
* Age >18
* Adequate organ function
* ECOG performance status < 3
* No prior therapies with selective inhibitors of mutated BRAF; other prior therapies must have been administered at least 4 weeks before administration of vemurafenib
* Life expectancy of at least 3 months
* Understanding and willingness to consent
* The use of corticosteroids to control cerebral edema or treat symptoms will be allowed
* A history of whole brain radiotherapy for brain metastases is allowed, but any stable lesion that was present at the time of WBRT will NOT be considered evaluable. A minimum of 1 week break will be required between prior WBRT and initiation of vemurafenib therapy.

Exclusion Criteria:

* Presence of leptomeningeal disease based on positive CSF cytology.
* History or presence of clinically significant ventricular or atrial dysrhythmias ≥ Grade 2 (NCI CTCAE, v4.0), Corrected QT (QTc) interval >450 ms at baseline or history of congenital long QT syndrome
* Uncontrolled medical illness, such as uncontrolled infection, congestive heart failure and MI within 2 months.
* Second active, untreated malignancy, which is likely to result in the patient's demise prior to death from uncontrolled melanoma CNS metastases. This will be determined on a case by case basis by the PIs.
* Unwillingness to undergo monitoring for a secondary malignancy including clinical dermatologic examinations and head and neck examinations and serial CT scans.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Harriet M Kluger, M.D., Principal Investigator — Yale University
Locations (1):
- Smilow Cancer Hospital at Yale New Haven, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vemurafenib Administration: Vemurafenib 960 mg orally, twice a day
Period: Overall Study
Arm/Group | Vemurafenib Administration
Started | 2
Completed | 0
Not Completed | 2
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Vemurafenib Administration
Number analyzed (Participants) | 2
Age, Continuous [Mean (Full Range); unit: years] | 42 [37 to 46]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Activity of Vemurafenib in Untreated Brain Metastases
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 1 year
Population: Subjects withdrew prior primary outcome measurement therefore no data was obtained to report
Arm/Group | Vemurafenib Administration
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event dating was collected through the duration of the study (approximately 14 months)
Arm/Group | Vemurafenib Administration
Serious Adverse Events (participants affected / at risk) | 1/2
Other Adverse Events (participants affected / at risk) | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vemurafenib Administration (N=2)
Nausea/Vomiting/Weakness (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes